CLINICAL TRIAL: NCT01191684
Title: A Phase I Study of an MVA Vaccine Targeting P53 in Cancer
Brief Title: Vaccine Therapy in Treating Patients With Colorectal, Stomach, or Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10105; NCI-2010-01859
Record Dates: First submitted 2010-08-27; First posted 2010-08-31 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Recurrent Colon Cancer; Recurrent Gastric Cancer; Recurrent Pancreatic Cancer; Recurrent Rectal Cancer; Stage III Colon Cancer; Stage III Gastric Cancer; Stage III Pancreatic Cancer; Stage III Rectal Cancer; Stage IV Colon Cancer; Stage IV Gastric Cancer; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms | interventions — Enzyme-Linked Immunosorbent Assay; Flow Cytometry; Immunoenzyme Techniques; MVAp53 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive MVAp53 subcutaneously on days 0, 21, and 42 in the absence of unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay; Other: flow cytometry; Other: immunoenzyme technique; Biological: modified vaccinia virus ankara vaccine expressing p53

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA
Other: flow cytometry — Correlative studies
Other: immunoenzyme technique — Correlative studies
  Other Names: immunoenzyme techniques
Biological: modified vaccinia virus ankara vaccine expressing p53 — Given SC
  Other Names: MVA-p53 vaccine; MVAp53 vaccine

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with colorectal, stomach, or pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:I. To establish whether 2 vaccine dose levels of modified vaccinia virus ankara vaccine expressing p53 (MVAp53) vaccines are safe and well tolerated in patients with p53 over-expressing solid tumor malignancy.

SECONDARY OBJECTIVES:I. To provide preliminary evidence of enhanced cellular and humoral immunity to p53.

OUTLINE:This is a phase I, dose-escalation trial of modified vaccinia virus ankara vaccine expressing p53 (MVAp53).Patients receive MVAp53 subcutaneously (SC) on days 0, 21, and 42 in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed up annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable and chemotherapy resistant primary or recurrent carcinoma of colorectal, gastric or pancreatic origin
* There must be pathologic evidence for malignancy with a soft tissue component of tumor evident on CT scan imaging or physical examination
* Patient must be able to give informed consent
* There must be an anticipated survival of at least 3 months
* Performance status of 80-100 (Karnofsky performance status)
* WBC count >= 3,000uL
* Platelet count >= 100,000uL
* Prothrombin time and partial thromboplastin time of <= 1.5 times the upper limit of normal
* Women of childbearing potential must have a negative pregnancy test; women and men of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant during or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Patients with asymptomatic small volume bone disease not likely to require radiation therapy during the period of the vaccine trial will be eligible
* Hemoglobin level > 9g/dL
* There must be evidence of p53 over expression by immunohistochemistry with > 10% of cells within the tumor strongly positive
* Patients with colorectal cancer will need to have failed to respond to 5-FU based therapy with oxaliplatin, irinotecan as well as epidermal growth factor receptor (EGFR) directed therapies (if appropriate); patients with gastric cancer will need to have progressed on standard first line chemotherapy or chemoradiotherapy and Herceptin based therapy (if appropriate); patients with pancreatic cancer who have failed to respond to at least 1 chemotherapy regimen

Exclusion Criteria:

* Diagnosis which has been associated with immunodeficiency, including HIV
* Prior radiation to more than 50% of all nodal groups
* Concurrent use of corticosteroids
* History of another malignancy, other than nonmelanoma skin cancer in the past 2 years
* Recent major surgery
* Serious intercurrent illness
* Temperature >= 101F within 3 days prior to the initial injection
* Pregnancy or lactation
* Clinically evident brain metastasis
* Autoimmune disease
* HIV seropositivity or refusal to hear the results of the HIV test
* Receipt of organ grafts
* History of severe environmental allergies
* History of severe neurological, cardiovascular, renal, hepatic, endocrine, respiratory, or bone marrow dysfunction requiring frequent re-evaluation, and management by a physician
* Patients with a history of congestive heart failure or coronary artery disease which has not been resolved by bypass or stent
* History of myopericarditis
* Known family history of Li-Fraumeni syndrome
* Allergy to egg proteins
* Chemotherapy or radiation within the 4 weeks preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance of modified vaccinia virus ankara vaccine expressing p53 assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4 toxicity scale | Assessed up to 12 months
  Safety data for each administered dose will be summarized using descriptive numbers and 95% confidence intervals from the exact binomial distributions

SECONDARY OUTCOMES:
Immunogenicity | Assesse up to 12 months
  Assessed using enzyme-linked immunosorbent assay (ELISA) for humoral response, lymphoproliferation for cluster of differentiation (CD)4+ T cell response, and intracytoplasmic cytokine assays, and interferon (IFN)-gamma and interleukin (IL)-4 by enzyme-linked immunosorbent spot (ELISPOT) for the assessment of cellular immune response. For each assay, the pre-vaccine values will be compared to the highest post-vaccine values. Immunogenicity changes and the maximum change will be quantified by mean, standard deviation, median, and range and tested by paired t-test at the 0.05 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Result] Hardwick NR, Carroll M, Kaltcheva T, Qian D, Lim D, Leong L, Chu P, Kim J, Chao J, Fakih M, Yen Y, Espenschied J, Ellenhorn JD, Diamond DJ, Chung V. p53MVA therapy in patients with refractory gastrointestinal malignancies elevates p53-specific CD8+ T-cell responses. Clin Cancer Res. 2014 Sep 1;20(17):4459-70. doi: 10.1158/1078-0432.CCR-13-3361. Epub 2014 Jul 1. PMID 24987057